CLINICAL TRIAL: NCT06392932
Title: Esophageal Temperature Dynamics and Injury During Pulmonary Vein Isolation With Temperature Controlled Very-High-Power Short-Duration Lesions Using the Novel Q-DOT Micro Ablation Catheter
Brief Title: Esophageal Temperature During PVI Using Q-DOT Micro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Eric Braunstein, Staff Physician I, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002707
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: Atrial Fibrillation; Esophageal thermal injury
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Prospective open-label randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Interpreters of the esophageal capsule endoscopy will be blinded to study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- QDOT Arm (Experimental): Temperature-controlled very-high-power short-duration ablation using the QDOT Micro catheter.
  Interventions: Device: QDOT Micro ablation catheter
- ST SF Arm (Active Comparator): Conventional high-power short-duration ablation using the ThermoCool ST SF catheter.
  Interventions: Device: ST SF ablation catheter

INTERVENTIONS:
Device: QDOT Micro ablation catheter — QDOT Micro ablation catheter
  Arms: QDOT Arm
Device: ST SF ablation catheter — ST SF ablation catheter
  Arms: ST SF Arm

SUMMARY:
This study will assess how two different ablation strategies, using two different ablation catheters during catheter ablation for paroxysmal atrial fibrillation, affect the temperature of the esophagus during ablation, and the risk of injury to the esophagus.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial, studying patients undergoing ablation involving pulmonary vein isolation for paroxysmal atrial fibrillation. Patients will be assigned to undergo conventional high-power short-duration ablation or temperature-controlled very-high-power short-duration ablation, and esophageal outcomes including temperature changes during ablation and esophageal injury as assessed by post-procedure capsule endoscopy will be compared between the groups. The hypothesis is that very-high-power short-duration ablation will lead to lower rises in esophageal temperature and lower rates of esophageal findings during capsule endoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged greater than or equal to 18 years
4. Diagnosed with paroxysmal atrial fibrillation
5. Undergoing RF catheter ablation for treatment of paroxysmal atrial fibrillation that will involve circumferential point-by-point radiofrequency ablation pulmonary vein isolation with no additional left atrial posterior wall ablation planned

Exclusion Criteria:

1. Patients who have undergone prior left atrial ablation procedures.
2. Patients where the use of the Q-DOT Micro ablation catheter in QMODE+ (i.e. temperature-controlled very-high-power short-duration ablation) is felt to be unsafe.
3. Patients who have contraindications to capsule endoscopy, or GI conditions that may increase the risks of capsule endoscopy (e.g. esophageal strictures, inflammatory bowel disease, etc)
4. Any records flagged "break the glass" or "research opt out."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Maximal change in esophageal temperature during posterior wall isolation. | During ablation procedure.

SECONDARY OUTCOMES:
Presence of esophageal thermal injury seen on post-procedure capsule endoscopy. | 2-4 days after ablation procedure.
Presence of procedural complications. | During and immediately following ablation procedure.

OTHER OUTCOMES:
Number of RF ablation lesions to performed pulmonary vein isolation. | During ablation procedure.
RF time during pulmonary vein isolation. | During ablation procedure.
Left atrial dwell time to achieve pulmonary vein isolation. | During ablation procedure.
Achievement of first pass pulmonary vein isolation. | During ablation procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Smidt Heart Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT06392932/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT06392932/ICF_001.pdf